CLINICAL TRIAL: NCT05481372
Title: Pioneering Imaging Techniques for Optimising Dose Delivery in Post-Operative Prostate Radiotherapy. A Feasibility Study.
Brief Title: PINPOINT Feasibility Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CCR 5380
Record Dates: First submitted 2022-07-28; First posted 2022-08-01 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Prostate Cancer; Image Guided Radiotherapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — X-Rays

STUDY DESIGN:
Intervention Model Description: Single centre feasibility study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Standard radiotherapy with research image acquisition (Experimental): Radiotherapy delivered as per standard of care Additional trans-perineal ultrasound (TPUS) imaging at three timepoints (1 x pre-treatment and 2 x treatment). Additional magnetic resonance imaging (MRI) pre-treatment.
  Interventions: Other: Imaging

INTERVENTIONS:
Other: Imaging — Trans-perineal ultrasound and Magnetic resonance image acquisition

SUMMARY:
This feasibility study is investigating the application of magnetic resonance imaging (MRI) and transperineal ultrasound (TPUS) to visualise potential sites of relapse and surrounding normal tissue in patient having post-operative prostate cancer radiotherapy. Structure visualisation on MRI and TPUS will be compared to current standard computer tomography (CT) and cone-beam computer tomography (CBCT) imaging.

DETAILED DESCRIPTION:
Approximately 47,000 men are diagnosed with prostate cancer yearly in the UK, 15% of which receive surgery (radical prostatectomy) as primary treatment. Of these men one third develop recurrence after prostatectomy and are offered post-operative radiotherapy.

Radiotherapy is targeted at the area where the prostate used to be, this includes potential relapse sites (PRS); vesicourethral anastomosis, bladder neck and retrovesicle space. When planning post-operative radiotherapy, the lack of a visible target means surrounding normal tissue is used to guide clinical target volume (CTV) delineation. The CTV is the area of tissue to be treated to the full radiotherapy prescription and includes PRS. Typically, the CTV is defined on a radiotherapy planning computer tomography (CT) scan.

The CTV lies adjacent to the bladder and rectum and is highly susceptible to positional changes influenced by organ filling. To identify and correct for CTV displacement during daily radiotherapy a cone-beam CT (CBCT) is acquired, this is an image similar to a CT scan but taken immediately prior to treatment delivery.

CT visualisation of PRS has been reported as inadequate, increasing the risk of missing or miss-identifying CTV structures during radiotherapy planning and delivery. To compensate for restricted visualisation on CT and CBCT an additional 1cm circumference around the CTV is treated to the prescription dose, this volume is referred to as the planning target volume (PTV). This margin reduces the risk of missing the target however its inclusion of normal tissue increases the risk of patient toxicity.

We propose that visualisation of PRS and surrounding normal tissue structures is enhanced on magnetic resonance imaging (MRI) compared to CT and on transperineal ultrasound (TPUS) compared to CBCT. This project investigates the reality of this statement by quantifying the confidence and reliability with which anatomical structures can be identified and delineated on all four image types.

ELIGIBILITY:
Inclusion Criteria:

* Patient has undergone radical prostatectomy
* Histologically confirmed prostate cancer
* Patient due to receive post-operative prostate bed +/- pelvic lymph node radiotherapy
* WHO performance status 0-1
* Age ≥ 18 years
* Written informed consent

Exclusion Criteria:

* Recruitment into POPS trial
* Contraindications to MRI such as having a pacemaker or non-MRI compatible implanted device

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Reliability of anatomical structure visualisation | 14 months
  Reliability of anatomical structure visualisation determined by mean dice similarity coefficient (DSC) and mean surface-to-surface distance (MSSD) for delineated structures (urethra, bladder neck, VUA, retrovesicle space, penile bulb, pubic symphysis and rectum) on MRI, CT, TPUS and CBCT across observers. If DSC is ≥ 0.75 the structure is deemed to be reliably visible.
Frequency of anatomical structure visualisation | 14 months
  Frequency of anatomical structure visualisation by average user rating of urethra, bladder neck, VUA, retrovesicle space, penile bulb, public symphysis and anterior rectal wall visualisation on MRI, CT, TPUS, CBCT and fused multimodality imaging (CT, MRI, TPUS).

SECONDARY OUTCOMES:
Anatomical structure motion | 14 months
  On TPUS, the distance (mm) between anterior rectal wall and posterior pubic symphysis measured every 30 seconds over 10 minutes and the distance (mm) between VUA and superior aspect of penile bulb measured every 30 seconds over 10 minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- Sophie Alexander, Sutton, Gastrointestinal (lower), United Kingdom

IPD SHARING:
Plan to Share IPD: No